CLINICAL TRIAL: NCT06999135
Title: Comparison of Silodosin and Tamsulosin for Medical Expulsive Therapy in Patients With Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Medical University (Other)
Responsible Party: Principal Investigator, DR FAIZA KHAN, ASSOCIATE PROFESSOR, Fatima Jinnah Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.31-Synopsis-FCPS-Pharma/FJ
Record Dates: First submitted 2025-04-17; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Tamsulosin; Silodosin; Medical Expulsive Therapy
MeSH Terms: interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAMSULOSIN (Active Comparator): Tamsulosin is an alpha-1 adrenergic receptor blocker commonly used to treat benign prostatic hyperplasia (BPH) by relaxing the smooth muscles in the prostate and bladder neck. In the context of medical expulsive therapy (MET), it helps facilitate the passage of ureteric stones by relaxing the smooth muscles of the lower ureter, reducing ureteric spasm, and easing stone expulsion. It is widely used due to its effectiveness and relatively well-tolerated side effect profile.
  Interventions: Drug: Silodosin
- Silodosin (Experimental): Silodosin is used as a medical expulsive therapy (MET) to facilitate the passage of distal ureteral stones, particularly those sized between 4 to 10 mm. It works by selectively blocking alpha-1A adrenergic receptors in the ureter, relaxing the smooth muscle, which helps stones pass more easily and quickly.
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — Silodosin is an oral medication primarily used to treat benign prostatic hyperplasia (BPH) by relaxing the muscles in the prostate and bladder neck to improve urine flow. It belongs to a class of drugs called alpha-1 adrenergic antagonists, which block receptors responsible for muscle contraction in these areas. This action helps relieve symptoms such as difficulty urinating, urgency, and weak urine stream. Silodosin is taken once daily with food and is known for its high selectivity for alpha-1A receptors, contributing to its effectiveness and safety profile
  Other Names: Sildat, Sildoso

SUMMARY:
This study compares the effectiveness and side effect profiles of Tamsulosin and Silodosin in medical expulsive therapy (MET) for ureteric stones. Conducted as a randomized control trial at Sir Ganga Ram Hospital, Lahore, 180 patients were analyzed-89 on Tamsulosin and 93 on Silodosin. Results showed that Silodosin had a higher stone expulsion rate, especially within 14 days, and fewer side effects compared to Tamsulosin. Common side effects included orthostatic hypotension, abnormal ejaculation, and headaches, with Silodosin showing a better overall safety profile.

DETAILED DESCRIPTION:
This study was designed as a prospective, randomized, open-label, controlled trial conducted at the Urology Department of Sir Ganga Ram Hospital, Lahore, over a period of 12 months. Ethical approval was obtained from the institutional review board, and written informed consent was secured from all participants.

Participants included adults aged 18 to 60 years with a single, unilateral ureteric stone measuring 5 to 10 mm, confirmed by non-contrast CT scan. Patients with a history of ureteral surgery, congenital anomalies, severe renal impairment (serum creatinine above 1.5 mg/dL), pregnancy, lactation, urinary tract infection, or those using calcium channel blockers or other alpha-blockers were excluded. A total of 180 eligible patients were randomized into two groups: 89 patients received Tamsulosin 0.4 mg daily, while 93 patients received Silodosin 8 mg daily.

Both groups received standard analgesia with diclofenac sodium 50 mg as needed and were advised to maintain adequate hydration. Treatment continued until stone expulsion or for a maximum of 28 days. Patients were monitored weekly through clinical evaluation and imaging (ultrasound or X-ray), and adverse events such as dizziness, ejaculatory dysfunction, and headaches were recorded using standardized questionnaires.

Data analysis was performed using SPSS version 25.0. Continuous variables were compared using Student's t-test, while categorical variables were assessed with Chi-square or Fisher's exact test. A p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages 18 years - 55 years.
* Solitary unilateral ureteral stone
* Stone sizes less than 10 mm measured on non-contrast computed tomography of kidney, ureter and bladder.
* Stones being treated primarily with medical expulsive therapy
* Radio opaque Stone

Exclusion Criteria:

* Pregnancy
* Untreated UTI
* Bleeding disorders
* Obstruction distal to stone
* Serum Creatinine > 1.3 mg/dl in males and > 1.2 mg/dl in females.
* Congenital renal anomaly/ skeletal malformation
* Previous treatment for the same stone (PCNL/ URS / push back)
* Solitary Kidney
* Prior JJ stent insertion
* Bilateral ureteral stone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
STONE EXPULSION RATE | 6 MONTHS
  This measure evaluates the proportion of patients who pass ureteral stones within specific time frames (0-14 days, 15-21 days, and 22-28 days) when treated with Silodosin versus Tamsulosin.
TIME TO STONE EXPULSION | 6MONTHS
  Number of days from treatment initiation to confirmed stone passage, measured by imaging and patient report.

SECONDARY OUTCOMES:
INCIDENCE OF ORTHOSTATIC HYPOTENSION | 6 months
  Percentage of patients experiencing orthostatic hypotension, measured by clinical blood pressure monitoring.
Incidence of Abnormal Ejaculation | 6 months
  Percentage of patients reporting abnormal ejaculation, assessed via patient questionnaires.
Incidence of Headache Percentage of patients reporting headaches, assessed via patient questionnaires. | 6 months
  Percentage of patients reporting headaches, assessed via patient questionnaires.
Analgesic Requirement: | 6 months
  Percentage of patients requiring analgesics during treatment, recorded from prescription or patient report.
Need for Auxiliary Procedures | 6 months
  Percentage of patients requiring interventions such as ureteroscopy or lithotripsy, documented from clinical records.
Stone Position and Laterality | 6 months
  : Distribution of stone location (proximal, mid, distal ureter) and side (right or left), determined by imaging.
Symptom Duration Prior to CT: | 6 months
  Categorized duration of symptoms before diagnosis, collected from patient history.

OTHER OUTCOMES:
BMI | 6 MONTHS
  Measurement: Categorized as Normal or Obese based on standard BMI thresholds (weight in kilograms divided by height in meters squared).

CONTACTS AND LOCATIONS:
Overall Officials: PROF MUNIZA QAYYUM, PHD PHARMACOLOGY, Study Chair — FATIMA JINNAH MEDICAL UNIVERSITY LAHORE
Locations (1):
- Fatima Jinnah Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Itoh Y, Okada A, Yasui T, Hamamoto S, Hirose M, Kojima Y, Tozawa K, Sasaki S, Kohri K. Efficacy of selective alpha1A adrenoceptor antagonist silodosin in the medical expulsive therapy for ureteral stones. Int J Urol. 2011 Sep;18(9):672-4. doi: 10.1111/j.1442-2042.2011.02810.x. Epub 2011 Jun 26. PMID 21707766
- [Background] Thongprayoon C, Krambeck AE, Rule AD. Determining the true burden of kidney stone disease. Nat Rev Nephrol. 2020 Dec;16(12):736-746. doi: 10.1038/s41581-020-0320-7. Epub 2020 Aug 4. PMID 32753740
- [Background] Kino M, Hayashi T, Hino D, Nakada T, Kitoh H, Akakura K. Patients' poor performance status is an independent risk factor for urosepsis induced by kidney and ureteral stones. Urolithiasis. 2021 Oct;49(5):477-484. doi: 10.1007/s00240-021-01256-4. Epub 2021 Mar 23. PMID 33755744
- [Background] 17. REHMAN I, KHAN H, FAROOQ A, MAHMOOD A, DIN QAM, HABIB B. Study on Uroliths Composition in Tertiary Care Hospital of Pakistan. Magnesium. 2021;7:18-9.
- [Background] Halinski A, Bhatti KH, Boeri L, Cloutier J, Davidoff K, Elqady A, Fryad G, Gadelmoula M, Hui H, Petkova K, Popov E, Rawa B, Saltirov I, Spivacow FR, Belthangady Monu Zeeshan Hameed, Trinchieri A, Buchholz N. Stone composition of renal stone formers from different global regions. Arch Ital Urol Androl. 2021 Oct 1;93(3):307-312. doi: 10.4081/aiua.2021.3.307. PMID 34839635
- [Background] Hsu YP, Hsu CW, Bai CH, Cheng SW, Chen KC, Chen C. Silodosin versus tamsulosin for medical expulsive treatment of ureteral stones: A systematic review and meta-analysis. PLoS One. 2018 Aug 28;13(8):e0203035. doi: 10.1371/journal.pone.0203035. eCollection 2018. PMID 30153301
- [Background] Rahman MJ, Faridi MS, Mibang N, Singh RS. Comparing tamsulosin, silodosin versus silodosin plus tadalafil as medical expulsive therapy for lower ureteric stones: A randomised trial. Arab J Urol. 2017 Dec 24;16(2):245-249. doi: 10.1016/j.aju.2017.11.012. eCollection 2018 Jun. PMID 29892490
- [Background] Sharma G, Pareek T, Kaundal P, Tyagi S, Singh S, Yashaswi T, Devan SK, Sharma AP. Comparison of efficacy of three commonly used alpha-blockers as medical expulsive therapy for distal ureter stones: A systematic review and network meta-analysis. Int Braz J Urol. 2022 Sep-Oct;48(5):742-759. doi: 10.1590/S1677-5538.IBJU.2020.0548. PMID 34003612
- [Background] Malin JM Jr, Deane RF, Boyarsky S. Characterisation of adrenergic receptors in human ureter. Br J Urol. 1970 Apr;42(2):171-4. doi: 10.1111/j.1464-410x.1970.tb10018.x. No abstract available. PMID 5420156
- [Background] Segura JW, Preminger GM, Assimos DG, Dretler SP, Kahn RI, Lingeman JE, Macaluso JN Jr. Ureteral Stones Clinical Guidelines Panel summary report on the management of ureteral calculi. The American Urological Association. J Urol. 1997 Nov;158(5):1915-21. doi: 10.1016/s0022-5347(01)64173-9. PMID 9334635
- [Background] Ibrahim AI, Shetty SD, Awad RM, Patel KP. Prognostic factors in the conservative treatment of ureteric stones. Br J Urol. 1991 Apr;67(4):358-61. doi: 10.1111/j.1464-410x.1991.tb15161.x. PMID 2032074
- [Background] Pietropaolo A, Proietti S, Geraghty R, Skolarikos A, Papatsoris A, Liatsikos E, Somani BK. Trends of 'urolithiasis: interventions, simulation, and laser technology' over the last 16 years (2000-2015) as published in the literature (PubMed): a systematic review from European section of Uro-technology (ESUT). World J Urol. 2017 Nov;35(11):1651-1658. doi: 10.1007/s00345-017-2055-z. Epub 2017 Jun 7. PMID 28593477
- [Background] Hughes T, Ho HC, Pietropaolo A, Somani BK. Guideline of guidelines for kidney and bladder stones. Turk J Urol. 2020 Nov;46(Supp. 1):S104-S112. doi: 10.5152/tud.2020.20315. Epub 2020 Oct 9. PMID 33052834
- [Background] Strohmaier WL, Wrobel BM, Schubert G. Overweight, insulin resistance and blood pressure (parameters of the metabolic syndrome) in uric acid urolithiasis. Urol Res. 2012 Apr;40(2):171-5. doi: 10.1007/s00240-011-0403-9. Epub 2011 Aug 25. PMID 21866382
- [Background] Ahmed AF, Al-Sayed AY. Tamsulosin versus Alfuzosin in the Treatment of Patients with Distal Ureteral Stones: Prospective, Randomized, Comparative Study. Korean J Urol. 2010 Mar;51(3):193-7. doi: 10.4111/kju.2010.51.3.193. Epub 2010 Mar 19. PMID 20414396
- [Result] Soliman MG, El-Gamal O, El-Gamal S, Abdel Raheem A, Abou-Ramadan A, El-Abd A. Silodosin versus Tamsulosin as Medical Expulsive Therapy for Children with Lower-Third Ureteric Stones: Prospective Randomized Placebo-Controlled Study. Urol Int. 2021;105(7-8):568-573. doi: 10.1159/000513074. Epub 2021 Feb 1. PMID 33524970
- [Result] Morita T, Wada I, Saeki H, Tsuchida S, Weiss RM. Ureteral urine transport: changes in bolus volume, peristaltic frequency, intraluminal pressure and volume of flow resulting from autonomic drugs. J Urol. 1987 Jan;137(1):132-5. doi: 10.1016/s0022-5347(17)43904-8. PMID 3795356

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT06999135/Prot_SAP_ICF_000.pdf